CLINICAL TRIAL: NCT01605838
Title: Pilot (Feasibility) Study of New Portable Monitor for Continuous Assessment of Cerebral Blood Flow (CBF) Autoregulation in Patients With Moderate to Severe Traumatic Brain Injury (TBI)
Brief Title: Noninvasive Monitoring of Cerebral Blood Flow Autoregulation in Patients With Traumatic Brain Injury (TBI)
Acronym: REG01
Status: Withdrawn | Type: Observational
Why Stopped: A series of administrative delays on all sides involved, combined with funding problems.
Sponsor: Advanced Brain Monitoring, Inc. (Industry)
Collaborators: University of Southern California (Other)
Responsible Party: Sponsor
Other Study IDs: ABM-TBI-0001; W81XWH - 10 - C - 0061 (Other Grant/Funding Number: DOD TATRC)
Record Dates: First submitted 2012-05-22; First posted 2012-05-25 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Traumatic Brain Injury (TBI)
Keywords: TBI
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
BACKGROUND: The brain is very sensitive to both excessive and insufficient flow of blood. Cerebral blood flow (CBF) is normally auto-regulated by the blood vessels in the brain, but this protective mechanism is often disturbed after a traumatic brain injury (TBI). Impairment or loss of the CBF autoregulation makes the brain vulnerable to oscillations of either arterial blood pressure (ABP) or intracranial pressure (ICP). The ideal management of TBI patients, therefore, involves continuous measurement and management of the cerebral perfusion pressure (CPP = ABP - ICP) but the measurement of CPP is currently possible only with specialized equipment and expertise that is not available in all institutions. The investigators have converted a no-longer used system that continuously monitors CBF autoregulation using rheoencephalography (REG) technology into a modern, small, battery-powered, low-cost monitor (aka BM-1) that acquires the REG signals using only noninvasive electrodes placed on the skin/scalp. REG data can then be used to calculate the optimal CPP to maintain in each individual patient. BM-1 is also capable of monitoring electroencephalography (EEG) and impedance plethysmography (IPG), which can, respectively, be used to measure brain electrical activity and changes in peripheral blood flow caused by blood pressure changes.

OBJECTIVES: The primary objectives are to (Obj. 1) demonstrate that REG acquired noninvasively is equal to the well-established but invasive method using intracranial pressure (ICP) monitoring, (Obj. 2) retrospectively test the idea that TBI patients have a less favorable outcome if their CPP were found less optimal using the REG data, and (Obj. 3) determine if noninvasive IPG or the PPG finger sensor monitoring (used to measure heart rate in doctor's offices) can replace the invasive monitoring of arterial blood pressure (ABP).

METHODOLOGY: This is an observational study with retrospective data analysis. 20 adult patients (18-65 yrs) with acute TBI, who meet the inclusion/exclusion criteria, will be enrolled on a first-come-first-enroll basis. The enrolled patients will have the REG, EEG and IPG signals monitored for the duration of ICU stay or 15 days, whichever is shorter. Standard neurological assessment will be made at the patient's discharge from the ICU and at 3 months after injury. The study is expected to end June 2013.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acute moderate or severe TBI
* Hospitalization within 12 hours from the injury
* Intraarterial catheterization and intracranial pressure (ICP) monitoring instantiated within 72 hours from the injury

Exclusion Criteria:

* Earlier head injuries, stroke, space-occupying intracranial lesions, meningitis, or cerebral vasculopathies
* Concomitant severe injuries of the chest, abdomen, pelvis, extremities or spine
* Concurrent terminal illness with a life expectancy of less than 6 months
* Unlikely to survive the next 48 hours after enrollment
* Implanted cardiac pacemaker, cardiac converter/defibrillator, or other electrical stimulator
* Pregnancy
* Patient is a prisoner or on a probation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (18 - 65 years) hospitalized in the surgical intensive care unit (ICU) because of moderate to severe traumatic brain injury
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-08; Primary Completion 2013-06 (Estimated); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Extended Glasgow Outcome Scale (GOSE) | 3 months post-injury

SECONDARY OUTCOMES:
Neurobehavioral Symptom Inventory (NSI) | 3 months post-injury
Rappaport Disability Rating Scale (DSR) | At discharge from intensive care unit; on average, 10 days post-injury
  Note regarding the time frame: based on the USC patient database for 2010 and 2011, patients may be discharged from the ICU anywhere between 4 days to 4 weeks; 50% of them will spend 10 +/- 3 days in the ICU.
Katz Index of Independence in Activities of Daily Living (KI-ADL) | 3 months post-injury

CONTACTS AND LOCATIONS:
Overall Officials: Djordje Popovic, MD, Principal Investigator — Advanced Brain Monitoring, Inc.
Locations (1):
- LA County + USC Medical Center, Los Angeles, California, United States

REFERENCES:
- [Background] Overgaard J, Tweed WA. Cerebral circulation after head injury. 1. Cerebral blood flow and its regulation after closed head injury with emphasis on clinical correlations. J Neurosurg. 1974 Nov;41(5):531-41. doi: 10.3171/jns.1974.41.5.0531. No abstract available. PMID 4418221
- [Background] Czosnyka M, Smielewski P, Kirkpatrick P, Menon DK, Pickard JD. Monitoring of cerebral autoregulation in head-injured patients. Stroke. 1996 Oct;27(10):1829-34. doi: 10.1161/01.str.27.10.1829. PMID 8841340
- [Background] Lam JM, Hsiang JN, Poon WS. Monitoring of autoregulation using laser Doppler flowmetry in patients with head injury. J Neurosurg. 1997 Mar;86(3):438-45. doi: 10.3171/jns.1997.86.3.0438. PMID 9046300
- [Background] Lang EW, Chesnut RM. A bedside method for investigating the integrity and critical thresholds of cerebral pressure autoregulation in severe traumatic brain injury patients. Br J Neurosurg. 2000 Apr;14(2):117-26. doi: 10.1080/02688690050004534. PMID 10889883
- [Background] Steiner LA, Czosnyka M, Piechnik SK, Smielewski P, Chatfield D, Menon DK, Pickard JD. Continuous monitoring of cerebrovascular pressure reactivity allows determination of optimal cerebral perfusion pressure in patients with traumatic brain injury. Crit Care Med. 2002 Apr;30(4):733-8. doi: 10.1097/00003246-200204000-00002. PMID 11940737
- [Background] Lang EW, Mehdorn HM, Dorsch NW, Czosnyka M. Continuous monitoring of cerebrovascular autoregulation: a validation study. J Neurol Neurosurg Psychiatry. 2002 May;72(5):583-6. doi: 10.1136/jnnp.72.5.583. PMID 11971041
- [Background] Schmidt B, Czosnyka M, Raabe A, Yahya H, Schwarze JJ, Sackerer D, Sander D, Klingelhofer J. Adaptive noninvasive assessment of intracranial pressure and cerebral autoregulation. Stroke. 2003 Jan;34(1):84-9. doi: 10.1161/01.str.0000047849.01376.ae. PMID 12511755
- [Background] Brady KM, Shaffner DH, Lee JK, Easley RB, Smielewski P, Czosnyka M, Jallo GI, Guerguerian AM. Continuous monitoring of cerebrovascular pressure reactivity after traumatic brain injury in children. Pediatrics. 2009 Dec;124(6):e1205-12. doi: 10.1542/peds.2009-0550. PMID 19948619
- [Background] Bodo M. Studies in rheoencephalography . Journal of Electrical Bioimpedance 2010; 1: 18 - 40.
- [Background] Bodo M, Pearce FJ, Montgomery LD, Rosenthal M, Kubinyi G, Thuroczy G, Braisted J, Forcino D, Morrissette C, Nagy I. Measurement of brain electrical impedance: animal studies in rheoencephalography. Aviat Space Environ Med. 2003 May;74(5):506-11. PMID 12751577
- [Background] Bodo M, Pearce FJ, Baranyi L, Armonda RA. Changes in the intracranial rheoencephalogram at lower limit of cerebral blood flow autoregulation. Physiol Meas. 2005 Apr;26(2):S1-17. doi: 10.1088/0967-3334/26/2/001. Epub 2005 Mar 29. PMID 15798222
- [Background] Bodo M, Pearce FJ, Armonda RA. Cerebrovascular reactivity: rat studies in rheoencephalography. Physiol Meas. 2004 Dec;25(6):1371-84. doi: 10.1088/0967-3334/25/6/003. PMID 15712716